CLINICAL TRIAL: NCT00698802
Title: Assessment of Safety and Efficacy of Biphasic Human Insulin IU 100 to EX1000 on Glycaemic Control in Subjects With Type 2 Diabetes
Brief Title: Safety and Efficacy of Biphasic Human Insulin Compared to EX1000 in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EX1000-1919
Record Dates: First submitted 2008-06-16; First posted 2008-06-17 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — biphasic human insulin 30

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: EX1000
- B (Active Comparator)
  Interventions: Drug: biphasic human insulin

INTERVENTIONS:
Drug: EX1000 — Treat-to-target titration scheme, s.c. injection
  Arms: A
Drug: biphasic human insulin — Treat-to-target titration scheme, s.c. injection
  Arms: B

SUMMARY:
This trial is conducted in Asia and Africa. This trial aims for a comparison of blood glucose control of biphasic human insulin 100 IU/mL and EX1000.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 12 months
* Current biphasic human insulin (BHI) for at least 3 months - as monotherapy or as the only insulin in combination with OADs
* Body Mass Index (BMI) less than or equal to 40.0 kg/m2
* HbA1c less than or equal to 9.5%
* FPG (SMPG) less than or equal to 12 mmol/L

Exclusion Criteria:

* Treatment with more than 1IU/kg insulin daily
* Treatment with Glucagon-like peptide 1 mimetics or dipeptityl peptidase IV inhibitors
* Known hypoglycaemia unawareness or recurrent major hypoglycaemia, as judged by the Investigator
* Known or suspected allergy to trial products or related products
* Receipt of any investigational drug within one month prior to this trial
* Any other condition that the Investigator feels would interfere with trial participation or evaluation of results, e.g. shiftworkers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 8 weeks of treatment

SECONDARY OUTCOMES:
HbA1c | For the duration of the trial
Fructosamine | For the duration of the trial
FPG | For the duration of the trial
4-point SMPG profiles | For the duration of the trial
Incidence of hypoglycaemic episodes | For the duration of the trial
Frequency and severity of adverse events (including injection site reactions) | For the duration of the trial
Laboratory safety parameters (haematology, biochemistry and lipids) | For the duration of the trial
Physical examination and vital signs | For the duration of the trial
Total daily insulin dosages | For the duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Vijayawada, India
- Johannesburg, Gauteng, South Africa
- Abu Dhabi, United Arab Emirates

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com